CLINICAL TRIAL: NCT05771883
Title: A Phase Ib/IIa Clinical Study of IMM0306 fo r Injection in Combination With Lenalidomide for the Treatment of Relapsed/Refractory CD20-Positive B-Cell Non-Hodgkin's Lymphoma Cell Non-Hodgkin's Lymphoma
Brief Title: A Clinical Study of Injectable IMM0306 in Combination With Lenalidomide
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM0306-003
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: B-cell Non-Hodgkin's Lymphoma
Keywords: 0306-03
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — Lenalidomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DLBCL and other B-NHL patients such as FL, MZL, MCL, etc. (Experimental): In this study, lenalidomide was administered at a fixed dose, in which 25 mg was used for DLBCL patients,and 20mg was used for other B-NHL patients such as FL, MZL, MCL, etc. and daily oral therapy with IMM0306 was used on the 1~21st day of each repeat 28-day cycle.
  The RP2D of the IMM0306 monotherapy trial was administered once a week (7 days ± 1 day) for intravenous infusion every 4 weeks
  Interventions: Drug: IMM0306; Drug: Lenalidomide capsule

INTERVENTIONS:
Drug: IMM0306 — IMM0306 is a fusion protein of CD20 mAb with the CD47 binding domain of SIRPα. The Fc segment of the recombinant protein in IMM0306 is IgG1 and has been modified by ADCC-enhanced genetic engineering.
  Other Names: IMM0306 Ingection
Drug: Lenalidomide capsule — Chemical name 3-(7-amino-3-oxo-1H-isoindol-2-yl)piperidin-2,6-dione, molecular formula C 13H 13 N 3 O 3, is an anti-tumor drug developed by Celgene Biopharmaceutical Company in the United States, with multiple effects such as anti-tumor, immunomodulatory and anti-angiogenesis
  Other Names: Revlimid

SUMMARY:
The objective of this study was to evaluate the safety and efficacy of IMM0306 in combination with lenalidomide in patients with relapsed/refractory CD20-positive B-cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
Main study purpose:

To assess the safety and tolerability of IMM0306 in combination with lenalidomide to determine the maximum tolerated dose (MTD) (if available) and the recommended Phase 2 dose (RP2D).

Secondary study purpose

1. To assess the antitumor efficacy of IMM0306 in combination with lenalidomide.
2. To assess the immunogenicity of IMM0306 in combination with lenalidomide.
3. To evaluate the pharmacokinetic (PK) profile of IMM0306 in combination with lenalidomide.

Exploratory study purpose:

1. Explore the correlation between exposure to IMM0306 and efficacy and safety (data permitting).
2. Explore the correlation of biomarkers with safety.

ELIGIBILITY:
Inclusion Criteria:

* 1)Patients should voluntarily sign the informed consent form, understand the study and be willing to follow the protocol and willing to complete all study procedures;
* 2)Male or female, aged ≥ 18 years old;
* 3)Phase Ib: CD20-positive B-cell non-Hodgkin lymphoma (B-NHL) diagnosed by histopathology which meets the criteria of 2016 WHO classification of lymphoid neoplasms, including but not limited to diffuse large B-cell lymphoma (DLBCL), follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone B-cell lymphoma (MZL), etc. Among them, indolent B-NHL must have failed at least 1 line of standard regimen, and aggressive B-NHL must have failed 2 or more lines of standard regimen. At least one regimen containing anti-CD20 monoclonal antibody monotherapy or in combination;

Phase IIa: CD20-positive B-cell non-Hodgkin lymphoma (B-NHL) of the following subtypes diagnosed by histopathology which meets the criteria of 2016 WHO classification of lymphoid neoplasms:

Cohort 1 Indications：Relapsed/refractory follicular lymphoma (FL, Grade 1-3a), 2 L； Inclusion Criteria：1）Histopathologically diagnosed CD20-positive FL Failure after first line treatment with regimens containing anti-CD20 monoclonal antibody monotherapy or in combination； Cohort 2 Indications：Relapsed/refractory marginal zone lymphoma (MZL), 2L

Classification of MZL:

* Splenic MZL
* Lymph node MZL Extramodal (MALT) Inclusion Criteria：1）Histopathologically diagnosed CD20-positive MZL Failure after first line treatment with regimens containing anti-CD20 monoclonal antibody monotherapy or in combination Cohort 3 Indications：Relapsed/refractory diffuse large B-cell lymphoma (DLBCL), 2 L Note: Including DLBCL transformed by follicular lymphoma Inclusion Criteria：1）Histopathologically diagnosed CD20-positive DLBCL Failure after first line treatment with regimens containing anti-CD20 monoclonal antibody monotherapy or in combination Note: Relapse is defined as disease progression after response (CR or PR) with adequate treatment, and at least one regimen containing anti-CD20; refractory is defined as failure to achieve a response after adequate treatment with regimen containing anti-CD20, or disease progression (PD or SD) during treatment/within 6 months after completion of adequate treatment.

Based on the safety and efficacy data from the Phase Ib study, the indications in the Phase IIa study may be adjusted, including the addition of new indications requiring determination of efficacy (eg, including but not limited to Waldenström's macroglobulinemia/lymphoplasmacytic lymphoma) or the deletion of indications (eg, including but not limited to DLBCL).

* 4)At least one measurable tumor lesion. Measurable lesions (2014 Lugano lymphoma response evaluation criteria (see details)): Longest diameter of lymph nodes > 15 mm, extranodal lesions > 10 mm; lesions previously treated with local therapy such as radiotherapy are considered measurable if disease progression has been demonstrated;
* 5)Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
* 6)Expected survival of at least 3 months;
* 7)The interval between the previous anti-tumor therapy and the first dose of this study must meet the following conditions: Prior anti-CD20 monoclonal antibody therapy with a discontinuation period of greater than 4 weeks; Prior CAR-T cell therapy with a washout period of greater than 4 weeks; Patients who have previously received chemotherapeutic drugs should discontinue for more than 4 weeks; Patients who have previously received small molecule targeted therapy should discontinue for more than 4 weeks; Patients who have previously received immune checkpoint inhibitors should discontinue for more than 8 weeks; Patients who have previously received surgery, radiotherapy and other anti-tumor drugs (including macromolecular targeted drugs, immunomodulators, traditional Chinese medicinal products with clear anti-tumor effect and indications of non-Hodgkin lymphoma, etc.) should have a interval of greater than 4 weeks;
* 8)Toxicities of prior anticancer therapy have been recovered to CTCAE v5.0 Grade ≤ 1 (except for residual alopecia effects) or baseline;
* 9)Adequate organ and hematopoietic function: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (no short-acting drugs for leucopenia within 1 week before the first dose and no long-acting drugs for leucopenia within 3 weeks before the first dose); Platelets ≥ 90 × 109/L (the patient has not received platelet transfusion therapy and thrombopoietin (TPO) therapy within 2 weeks before the first dose); Hemoglobin ≥ 90 g/L (patient has not received red blood cell transfusion therapy or erythropoietin (EPO) therapy within 2 weeks prior to the first dose); Serum creatinine (formula is shown in 附录 2) ≤ 1.5 times of upper limit of normal (ULN) or endogenous creatinine clearance (CCr) ≥ 50 mL/min; for subjects with urine protein ≥ 2 + detected by urine dipstick at baseline, 24-hour urine protein quantitative test shall be performed, and the result shall be < 1g; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 times ULN for patients without liver involvement; AST and ALT ≤ 5.0 times ULN for patients with liver involvement; Serum total bilirubin (TBIL) ≤ 1.5 times ULN; International normalized ratio (INR) ≤ 2 times ULN, or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;
* 10)Female patients of childbearing potential must have a negative blood pregnancy test within 7 days prior to the first dose; any male and female patients of childbearing potential must agree to use an effective method of contraception throughout the study and for 6 months after the last dose of study drug. (Details are shown in Appendix 7)

Exclusion Criteria:

* 1)Patients with current or previous primary central nervous system lymphoma (PCNSL) or secondary central nervous system involvement. Patients with central nervous system symptoms must undergo lumbar puncture and magnetic resonance imaging (MRI) for exclusion;
* 2)Patients who have received allogeneic hematopoietic stem cell transplant or other organ transplant or received autologous hematopoietic stem cell transplant within 100 days prior to the first dose;
* 3)Patients who have received live attenuated vaccines within 4 weeks prior to the first dose or planned during the study;
* 4)Patients with a history of malignancy within the last 5 years, except for patients with completely cured basal cell carcinoma of skin or squamous cell carcinoma of skin, melanoma in situ, and cervical carcinoma in situ and/or patients with any malignancy for whom the cancer has been cured without disease or for at least 5 consecutive years without disease;
* 5)Patients with active autoimmune diseases or medical history that may relapse (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disorder, multiple sclerosis, vasculitis, glomerulonephritis, etc.), or patients at high risk. However, the following patients may be considered for enrollment if they have stable disease as assessed by the investigator: Autoimmune hypothyroidism requiring only hormone replacement therapy; Skin disease not requiring systemic treatment (e.g., eczema, rash accounting for less than 10% of the body surface);
* 6)Patients who have undergone major surgery within 28 days prior to the first dose or are expected to have major surgery during this study;
* 7)Subjects with deep venous embolism or pulmonary artery embolism within 6 months prior to screening;
* 8)Subjects requiring treatment with systemic corticosteroids (> 10 mg/day prednisone or equivalent dose) or other immunosuppressive agents within 7 days prior to the first dose or during the study, except for topical glucocorticoids administered by nasal spray, inhalation, or other routes, or physiological doses of systemic glucocorticoids;
* 9)Patients who require chronic oral administration of aspirin or other non-steroidal anti-inflammatory drugs, clopidogrel and other drugs that inhibit platelet aggregation (except for patients who meet the inclusion criteria who can suspend the treatment as assessed by the investigator);
* 10)Patients with current interstitial lung disease or pneumonitis, active tuberculosis infection;
* 11)Patients with systemic diseases not stably controlled after treatment, such as diabetes, severe organic cardiovascular and cerebrovascular diseases;
* 12)The patient's heart meets any of the following conditions: Left ventricular ejection fraction (LVEF) ≤ 55%; Congestive heart failure or active heart disease of New York Heart Association (NYHA) (see Appendix 3) Class II or greater; Serious arrhythmia requiring treatment (except for atrial fibrillation and paroxysmal supraventricular tachycardia which are judged by the investigator as having no effect on the study); QTc interval ≥ 450 ms for males and ≥ 470 ms for females (QTc formula is shown in Appendix 4); Have myocardial infarction or bypass or stent surgery within 6 months before administration; Other cardiac diseases that are not suitable for enrollment judged by the investigator;
* 13)Patients with human immunodeficiency virus (HIV) infection, hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) positive at screening, and HBV-DNA above the lower limit of measurement; HCV antibody positive at screening and HCV-RNA above the lower limit of measurement;
* 14)Evidence of uncontrollable serious active infection at screening (eg, sepsis, bacteremia, fungemia, viremia, etc);
* 15)Subjects with known previous severe allergic reactions (CTCAE v5.0 grade ≥ 3) to macromolecular protein preparations/monoclonal antibodies and any components of the investigational product;
* 16)Subjects who have participated in other interventional drug or medical device clinical studies or are receiving other clinical study treatments (other than non-interventional studies) within 4 weeks prior to the first dose of this study;
* 17)Patients with a clear past history of neurological or mental disorders, such as epilepsy, dementia, and poor compliance;
* 18)Pregnant or lactating women;
* 19)Patients with history of stroke or intracranial hemorrhage within 6 months;
* 20)Patients with active or documented haemorrhage of digestive tract within 6 months (eg, esophageal or gastric varices, ulcer bleeding);
* 21)Patients who are ineligible for participation in this study in the opinion of the investigator for other reasons, such as rapid disease progression at screening, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Though end of DLT evaluation period,up to approximately 28 days.
  To be summarized using descriptive statistics
Maximum Tolerated Dose (MTD) | Dose-limiting toxicities will be evaluated during the first cycle (28 days) of treatment.
  If the planned dose escalation of IMM0306 in combination with lenalidomide to a preset highest dose group (i.e., the single-agent RP2D dose recommended in the IMM0306-I trial) does not reach MTD, it will be possible to continue to increase the dose exploration or explore new frequency of administration. SMC will also review pre-safety data and recommend whether to further increase the dose and explore new dosing frequencies.